CLINICAL TRIAL: NCT05380830
Title: Metabolic Alterations in Obese Women Undergoing High-intensity Physical Exercise Associated With Intermittent Recovery Hypoxia.
Brief Title: Metabolism of Obese Women Under Exercise and Recovery Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DWR_Hypoxia
Record Dates: First submitted 2022-05-07; First posted 2022-05-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity; Intermittent hypoxia; Metabolic disease; Deep-water running
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
Who Masked: Participant
Masking Description: Participants will be randomly distributed into 3 groups: Control (Gcon), Hypoxia (GHyp) and Normoxia (GNor). Those in Ghyp and GNor won't be able to know which group they are.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The group will be only submitted to evaluations (body composition, hematological, lipid and cytokines profile, food intake, and maximal effort under treadmill and deep-water running) at the beginning and the end of the study.
- Group Hypoxia (Experimental): During the intervention of 8 weeks the participants will have the deep-water running training under normoxia, but during the rest they will be under hypoxia (FiO2=13%).
  Interventions: Other: Tied deep-Water Running
- Group Normoxia (Placebo Comparator): During the intervention of 8 weeks the participants will have the deep-water running training under normoxia, and during the rest they will keep under normoxia (FiO2=20%).
  Interventions: Other: Tied deep-Water Running

INTERVENTIONS:
Other: Tied deep-Water Running — 4 efforts of tied deep-water running for 5 minutes at 100-110%Vo2max under normoxia with 5 minutes of passive rest under hypoxia (FiO2=13%) or normoxia (FiO2= 20%). Frequency: 3x/week for 8 weeks.
  Other Names: DWR
  Arms: Group Hypoxia; Group Normoxia

SUMMARY:
Obesity is characterized as a low-grade systemic inflammatory disease, which changes several pro-and anti-inflammatory cytokines. The practice of physical activity is a non-pharmacological method that results in the reduction of the systemic inflammatory state and, when associated with hypoxia exposure, may substantially improve this state. Deep-water running is highly indicated to obese for guarantee less joint impact and lower fatigue levels. In this way, the high-intensity exercise associated with intermittent recovery hypoxia in obese women will be investigated.

DETAILED DESCRIPTION:
Obesity is characterized as a low-grade systemic inflammatory disease. With the increase in adipose tissue, several cytokines show alterations in synthesis and secretion, resulting in endocrine imbalances. The cytokines that most influence this process are adiponectin, which is anti-inflammatory and reduces its concentration during obesity. At the same time, the pro-inflammatory cytokines are tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6), which show a significant increase in the face of obesity. The practice of physical activity is a non-pharmacological method that results in the reduction of the systemic inflammatory state, altering the lipid profile and levels of both anti- and pro-inflammatory cytokines and the improvement of the individual's physical capacity. Due to the high joint overload and muscle stress, water exercises are recommended for obese individuals as it maintains motor stimulation with a low risk of injury. The training tied to running in a deep pool, also known as Deep Water Running (DWR), will promote advantages similar to running on the ground, such as improving aerobic capacity, avoiding impact and enabling the performance of exercise at high intensities lower levels of fatigue. The high-intensity exercise performance reduces the availability of oxygen to muscle cells, inducing the hypoxic environment, which causes stabilization of the hypoxia inductive factor 1 (HIF-1), promoting gene transcriptions related to erythropoiesis and angiogenesis. Thus, the present study aims to investigate the effects of high-intensity physical exercise associated with recovery hypoxia, observing both the inflammatory and lipid profile and the physical capacity of obese women grade I. For this, 45 women with obesity will participate in the study, divided into 3 groups: hypoxia, normoxia and control. All will perform body composition, food intake, hematological and lipid profile tests, plus the serum quantification of cytokines before and after the 8 weeks of physical training. Deep-water tied running (DWR) training will be periodized, high-intensity interval, with recovery in hypoxia or normoxia. Intermittent recovery hypoxia is expected to act as an additive effect on the use of oxygen by the muscle, resulting in an improvement in the hematological and lipid profile, aerobic capacity and changes in the inflammatory profile in obese women.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age between 25 - 45 years old;
* BMI between 30 - 35kg/m²;
* Not be on a diet;
* Not be on a physical activity program;
* Not be menopaused.

Exclusion Criteria:

* Smokers;
* Alcoholics;
* Use thyroid medication;
* Carry out nutritional monitoring or in treatment for weight loss;
* Hypertension;
* Metabolical syndrome;
* Have any comorbidity associated to obesity;
* Drugs use.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Body weight changes (Anthropometry) | Eight weeks
  Changes in body weight (kilograms - Kg) pre- and post- intervention.
Height assessment (Anthropometry) | Eight weeks
  Height measured in meters
Body mass index changes (Anthropometry) | Eight weeks
  Changes in body mass index (BMI = weight measured(kg) / (height (m)²) evaluated pre- and post- intervention.
Body composition changes (Anthropometry) | Eight weeks
  Changes in fat-free mass, fat mass and bone mineral content evaluated pre- and post- intervention. Dual energy x-ray absorptiometry (DEXA) will be use.
Erythrogram (Hematological profile) | Eight weeks
  The red cells, hematocrit cells and hemoglobin will be evaluated pré- and post- intervention using a Radiometer-ABL 700 (Radiometer, Copenhagen, Denmark), and for erythropoietin evaluation an EPO Immunoassay ELISA kit will be used.
EPO (Hematological profile) | Eight weeks
  The erythropoietin will be evaluated with an EPO Immunoassay ELISA kit in pre- and post- intervention .
Lipid profile | Eight weeks
  Changes in total cholesterol, triglycerides, HDL-cholesterol and LDL-cholesterol and blood glucose evaluated pre- and post- intervention, quantified by Total Liquiform Cholesterol Kit, HDL Cholesterol Kit and Liquiform Triglycerides Kit, from Labtest diagnóstica®, using an enzymatic system and absorbance spectrophotometer.
Inflammatory profile | Eight weeks
  Changes in serum levels of cytokines IL-6, TNF-α, adiponectin, FBP4 and leptin will be evaluated pre- and post- intervention, by MILLIPLEX® Kit.
Changes in aerobic performance (deep-water running) | eight weeks
  Physical tests performed pre-, after 4 weeks and post- intervention to assess aerobic physical fitness by incremental test in treadmill. The test aim to evaluate the anaerobic threshold (AT) and VO2peak in deep-water running.
Changes in aerobic performance (treadmill) | eight weeks
  Physical tests performed pre-, after 4 weeks and post- intervention to assess aerobic physical fitness by incremental test in treadmill. The test aim to evaluate the anaerobic threshold (AT) and VO2peak in treadmill.
Food Intake changes | Eight weeks
  A food record of three non-consecutive days: two days of the week and one day in the weekend. This evaluation will last eight weeks. The caloric intake, macronutrients and fiber will be evaluated over the intervention with Dietwin® software (São Paulo, Brazil).
Processed and ultraprocessed food intake changes | Eight weeks
  The feed will undergo analysis through the NOVA Classification. By NOVA, food will be classified into four groups: Group 1 - Unprocessed or minimally processed foods; Group 2 - Processed culinary ingredients; Group 3 - Processed foods; Group 4 - Ultra-processed foods. For each category, the total calories ingested will be calculated, and later, represented in percentage (%) the participation of each food group in the general diet.

SECONDARY OUTCOMES:
Rate of Perceived Effort (RPE) | eight weeks
  The rate of perceived effort (RPE) will be noted after each effort during all the training program. The Borg scale will be used.
Oxygen saturation (SpO2) | Eight weeks
  For group hypoxia and normoxia the oxigen saturation will be followed during the rest with a pulse oximeter. The SpO2 will be noted after the end of the effort, after 2,5 minutes in rest and in the end of the rest.
Internal load (TRIMP) | Eight weeks
  The .internal load will be calculated using TRIMP, that is calculated multipling the RPE for the time in effort (TRIMP = RPE * time in effort), for each participant and training session.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela C Lima Viliod, Principal Investigator — USP
Locations (1):
- University of São Paulo, School of Physical Education and Sports of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No